CLINICAL TRIAL: NCT01646268
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study Of The Efficacy And Safety Of The Rotigotine Transdermal Patch In Chinese Subjects With Early-stage Idiopathic Parkinson's Disease
Brief Title: Rotigotine Versus Placebo As Double Blind Study To Evaluate The Efficacy In Early Stage Idiopathic Parkinson's Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0914
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: IDIOPATHIC PARKINSON'S DISEASE
Keywords: Rotigotine; Neupro phase 3; Early phase; Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): Rotigotine, daily doses, treatment group
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Placebo, daily doses, placebo group
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Rotigotine — Transdermal Patch
  Content:
  2 mg /24 h (10 cm^2), 4 mg /24 h (20 cm^2), 6 mg /24 h (30 cm^2), 8 mg /24 h (40 cm^2)
  For early-stage Parkinson's disease, receive Rotigotine patches in escalating weekly dose (starting with daily doses 2 mg/24 h to 8 mg/24 h) for a maximum 4-week Titration Period, then 24 week maintenance period
  Arms: Rotigotine
Drug: Placebo Patch — Transdermal Patch
  Size:
  10 cm^2, 20 cm^2, 30 cm^2, 40 cm^2
  Subjects randomized to placebo will receive matching placebo patches
  Arms: Placebo

SUMMARY:
The primary objective is to demonstrate that the Rotigotine transdermal patch is efficacious in Chinese subjects with early-stage idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
The study includes a maximum 4-week Screening Period, a maximum 4-week Titration Period for early-stage Parkinson's disease 24-week Maintenance Period, a maximum 6-day De-escalation Period and 30-day Safety Follow-Up Period. The maximum study durations for an individual subject with early-stage Parkinson's disease will be 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* An Independent Ethics Committee (IEC)-approved written informed consent is signed and dated by the subject or by the legal representative
* Subject/legal representative is considered reliable and capable of adhering to the protocol, visit schedule or study medication intake according to the judgment of the investigator
* Subject has Idiopathic Parkinson's Disease of ≤5 years' duration, defined by the cardinal sign, Bradykinesia, plus the presence of at least 1 of the following: resting tremor, rigidity, or impairment of postural reflexes, and without any other known or suspected cause of Parkinsonism
* Subject is Hoehn & Yahr stage ≤3
* Subject is male or female aged ≥30 years at Screening (Visit 1)
* Subject has a Mini Mental State Examination (MMSE) score of ≥25
* Subject has a Unified Parkinson's Disease Rating Scale (UPDRS) motor score (Part III) of ≥10 at Baseline (Visit 2)
* If the subject is receiving an Anticholinergic agent (eg, Benztropine, Trihexyphenidyl, Parsitan, Procyclidine, Biperiden), a monoamine oxidase (MAO)-B inhibitor (eg, Selegiline), an N-methyl-d-aspartate (NMDA) antagonist (eg, Amantadine), he/she must have been on a stable dose for at least 28 days prior to Baseline (Visit 2) and be maintained on that dose for the duration of the study

Exclusion Criteria:

* Subject has previously participated in this study or subject has previously received the study medication under investigation in this study
* Subject is participating in another study of an investigational drug or has done so within 28 days prior to the Baseline Visit (Visit 2)
* Subject has a history of significant skin hypersensitivity to adhesive or other transdermal preparations or recent unresolved contact Dermatitis
* Subject has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening (Visit 1)
* Subject has atypical Parkinson's syndrome(s) due to drugs (eg, Metoclopramide, Flunarizine), metabolic neurogenetic disorders (eg, Wilson's Disease), Encephalitis, Cerebrovascular Disease, or Degenerative Disease (eg, progressive Supranuclear Palsy)
* Subject has a history of Pallidotomy, Thalamotomy, deep brain stimulation, or fetal tissue transplant
* Subject has dementia, active psychosis or hallucinations, or severe depression
* Subject is receiving therapy with a dopamine agonist either concurrently or has done so within 28 days prior to the Baseline Visit (Visit 2)
* Subject is receiving therapy with L dopa/carbidopa and/or L-dopa/benserazide within 28 days of Baseline (Visit 2) or has received L-dopa/carbidopa and/or L-dopa/benserazide for more than 6 months since diagnosis
* Subject is receiving therapy with 1 of the following drugs either concurrently or within 28 days prior to Baseline (Visit 2): Alpha-methyl dopa, Metoclopramide, Reserpine, Neuroleptics (except specific atypical neuroleptics: Olanzapine, Ziprasidone, Aripiprazole, Clozapine, Quetiapine), MAO-A inhibitors, Methylphenidate, or Amphetamine
* Subject is currently receiving central nervous system (CNS) active therapy (eg, sedatives, hypnotics, antidepressants, anxiolytics), unless the dose has been stable for at least 28 days prior to Baseline Visit (Visit 2) and is likely to remain stable for the duration of the study
* Subject has a current diagnosis of Epilepsy, has a history of seizures as an adult, has a history of stroke, or has had a transient ischemic attack within 1 year prior to Screening (Visit 1)
* Subject has clinically relevant hepatic dysfunction (as defined as a total bilirubin >2.0 mg/dL or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than 2 times the upper limit of the reference range)
* Subject has clinically relevant renal dysfunction (serum creatinine >2.0 mg/dL [>178 umol/L])
* Subject has clinically relevant cardiac dysfunction (any cardiac disorder which in the opinion of the investigator would put the subject at risk of clinically relevant arrhythmia) and/or myocardial infarction within the last 12 months
* Subject has a QT interval corrected for heart rate according to Bazett's formula (QTcB) of ≥500 ms at Screening (Visit 1)
* Subject has a history of only symptomatic (not asymptomatic) orthostatic hypotension with a decrease of systolic blood pressure (SBP) from supine to standing position of ≥20 mmHg or of ≥10 mmHg in diastolic blood pressure (DBP) after 1 or 3 minutes within 28 days prior to the Baseline Visit (Visit 2), or SBP less than 105 mmHg at study entry
* Subject has evidence of an impulse control disorder (ICD) at Screening (Visit 1)
* Subject has a history of known intolerance/hypersensitivity to the following Antiemetics; Domperidone, Trimethobenzamide, Ondansetron, Tropisetron, Granisetron, and Glycopyrrolate
* Subject has a history of chronic alcohol or drug abuse within the last 5 years
* Subject is pregnant or nursing, or is of childbearing potential but (i) not surgically sterile or (ii) not using adequate birth control methods (including at least a double barrier method) or (iii) not sexually abstinent or (iv) not at least 2 years post-menopausal
* Subject has any other clinically relevant medical condition, psychiatric condition, or laboratory abnormality, which would in the judgment of the investigator, interfere with the subject's ability to participate in the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 1 877 822 9493
Locations (24):
- China (24):
  - 001, Beijing
  - 002, Beijing
  - 019, Beijing
  - 025, Beijing
  - 017, Changchun
  - 007, Chengdu
  - 027, Chengdu
  - 021, Fuzhou
  - 010, Guangzhou
  - 011, Guangzhou
  - 014, Guangzhou
  - 015, Guangzhou
  - 005, Hangzhou
  - 013, Hangzhou
  - 018, Hangzhou
  - 023, Jinan
  - 003, Shanghai
  - 004, Shanghai
  - 009, Shanghai
  - 008, Suzhou
  - 016, Tianjin
  - 006, Wuhan
  - 022, Wuhan
  - 024, Wuhan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The SP0914 study began recruitment in July 2012 and concluded in May 2014. All subjects were recruited in China.
Pre-assignment Details: The Participant Flow and Demographics data is taken from the Randomized Set (RS). The RS includes all subjects that were randomized.
Groups:
- Rotigotine: Rotigotine, daily doses, treatment group
  Rotigotine: Transdermal Patch
  Content:
  2 mg /24 h (10 cm^2), 4 mg /24 h (20 cm^2), 6 mg /24 h (30 cm^2), 8 mg /24 h (40 cm^2)
  For early-stage Parkinson's disease, receive Rotigotine patches in escalating weekly dose (starting with daily doses 2 mg/24 h to 8 mg/24 h) for a maximum 4-week Titration Period, then 24 week maintenance period.
- Placebo: Placebo, daily doses, placebo group
  Placebo Patch: Transdermal Patch
  Size:
  10 cm^2, 20 cm^2, 30 cm^2, 40 cm^2
  Subjects randomized to placebo will receive matching placebo patches.
Period: Overall Study
Arm/Group | Rotigotine | Placebo
Started | 124 | 123
Completed | 113 | 107
Not Completed | 11 | 16
Not completed — Adverse Event | 6 | 7
Not completed — Lack of Efficacy | 1 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Demographics data is taken from the Randomized Set (RS). The RS includes all subjects that were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotigotine | Placebo | Total
Number analyzed (Participants) | 124 | 123 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 82 | 170
  >=65 years | 36 | 41 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.3) | 59.7 (10.1) | 59.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 97
  Male | 74 | 76 | 150
Region of Enrollment [Number; unit: participants]
  China | 124 | 123 | 247
Weight [Mean (Standard Deviation); unit: kilograms] | 63.2 (10.5) | 64.0 (9.9) | 63.6 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Sum of the Score From the Activities of Daily Living (ADL) Scale and Motor Examination in the Unified Parkinson's Disease Rating Scale (UPDRS) (Parts II+III, a UPDRS Subtotal) From Baseline to the End of Double-blind Maintenance Period
Description: The UPDRS assessments (Parts II+III) will be performed at every visit.
  For the assessment of the subject's disability, Part II of the UPDRS will be used. Data will be gathered pertaining to the subject's disease state in the "on" state. Subjects will respond to questions about their general state in the week prior to their scheduled visit in conjunction with any observations made by the investigator (or designee). For the assessment of the subject's motor function, Part III of the UPDRS will be used and the assessments will be done while the subject is in the "on" state.
  The UPDRS Part II (Activities of Daily Living) consists of 13 items scored between 0 and 4. The UPDRS Part III (motor subscale) consists of 27 items and sub items scored between 0 and 4. The sum score is calculated as sum of these 27 individual scores. The sum score ranges from 0 to 160, higher scores denote greater disability.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 24)
Population: This analysis consists of the Full Analysis Set [Last Observation Carried Forward], which includes all subjects who are randomized, receive at least 1 dose of study medication, and have a Baseline efficacy measurement and at least 1 post-Baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 123 | 121
units on a scale | -4.9 (9.9) | -0.2 (9.9)
Statistical Analysis 1: Comparison: Rotigotine vs Placebo; The null hypothesis (H0) is that there is no difference in the change in the sum of the score from the ADL and motor examination in the UPDRS (Parts II+II) between the active treatment and the placebo groups (i.e., the change from Baseline in the sum of the score from the ADL and motor examination in the UPDRS (Parts II+III) is the same for both groups); Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Means = -4.82, 95% CI 2-sided [-7.18 to -2.45], Standard Error of Mean 1.20 — Value describes the difference value of the mean change from baseline between Rotigotine and Placebo groups. The Value for this outcome was -4.6

2. Secondary Outcome: Response to Therapy, Defined as ≥20 % Decrease in the Sum of Scores From Activities of Daily Living (ADL) & Motor Examination in Unified Parkinson's Disease Rating Scale (UPDRS Parts II+III, a UPDRS Subtotal) From Baseline to End of Maintenance Period
Description: The UPDRS assessments (Parts II+III) will be performed at every visit. For the assessment of the subject's disability, Part II of the UPDRS will be used. Data will be gathered pertaining to the subject's disease state in the "on" state. Subjects will respond to questions about their general state in the week prior to their scheduled visit in conjunction with any observations made by the investigator (or designee). For the assessment of the subject's motor function, Part III of the UPDRS will be used and the assessments will be done while the subject is in the "on" state.
  The UPDRS Part II (Activities of Daily Living) consists of 13 items scored between 0 and 4. The UPDRS Part III (motor subscale) consists of 27 items and sub items scored between 0 and 4. The sum score is calculated as sum of these 27 individual scores. A higher score denotes greater disability.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 24)
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 123 | 121
percentage of responders | 42.3 | 22.3

3. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale [UPDRS Part II (ADL)] From Baseline to the End of the Double-blind Maintenance Period
Description: The UPDRS assessments (Parts II+III) will be performed at every visit.
  For the assessment of the subject's disability, Part II of the UPDRS will be used. Data will be gathered pertaining to the subject's disease state in the "on" state. Subjects will respond to questions about their general state in the week prior to their scheduled visit in conjunction with any observations made by the investigator (or designee). The UPDRS Part II (Activities of Daily Living) consists of 13 items scored between 0 and 4. The sum score ranges from 0 to 52, higher scores denote greater disability.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 123 | 121
units on a scale | -1.4 (3.6) | 0.1 (3.4)

4. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale [UPDRS Part III (Motor Examination)] From Baseline to the End of the Double-blind Maintenance Period
Description: The UPDRS assessments (Parts II+III) will be performed at every visit.
  For the assessment of the subject's motor function, Part III of the UPDRS will be used and the assessments will be done while the subject is in the "on" state.
  The UPDRS Part III (motor subscale) consists of 27 items and sub items scored between 0 and 4. The sum score ranges from 0 to 108, higher scores denote greater disability.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 123 | 121
units on a scale | -3.4 (7.3) | -0.3 (7.4)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected throughout the duration of the SP0914 study (approximately 2 years). AE data consists of the Safety Set (SS). The SS includes all randomized subjects who received at least 1 dose of study medication.
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
  AE and SAE data represents Treatment-emergent Adverse Events (TEAE).
Arm/Group | Rotigotine | Placebo
Serious Adverse Events (participants affected / at risk) | 6/124 | 1/123
Other Adverse Events (participants affected / at risk) | 35/124 | 18/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=124) | Placebo (N=123)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial bridging (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=124) | Placebo (N=123)
Nausea (Gastrointestinal disorders) | 11 (16) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (9) | 2 (2)
Somnolence (Nervous system disorders) | 10 (10) | 4 (4)
Dizziness (Nervous system disorders) | 10 (13) | 7 (9)
Erythema (Skin and subcutaneous tissue disorders) | 8 (11) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (12) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.